CLINICAL TRIAL: NCT00339625
Title: Polyp Prevention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9999910159; OH91-C-0159
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Diet; Polyps; Adenoma
Keywords: Intervention; Diet; Colon
MeSH Terms: conditions — Polyps; Adenoma | interventions — Diet, Fat-Restricted

ARMS (2):
- 1 (Experimental): low fat, high fiber, high fruit and vegetable eating plan
  Interventions: Other: low fat, high fiber, high fruit and vegetable eating plan
- 2 (No Intervention): Usual Diet

INTERVENTIONS:
Other: low fat, high fiber, high fruit and vegetable eating plan — Participants were randomized to a low fat, high fiber, high fruit and vegetable (intervention arm) or their usual diet (control arm)
  Arms: 1

SUMMARY:
The primary objective of the Poly Prevention Trial (PPT) is to determine whether a low fat, high fiber, high vegetable and fruit eating plan will decrease the recurrence of adenomatous polyps of the large bowel. Secondary objectives of the PPT include 1) evaluating the effectiveness of the intervention program with respect to participant achievement of dietary goals; 2) examining the relation of dietary change and biochemical markers in blood; and 3) assessing the impact of the intervention on quality of life indicators.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective of the Polyp Prevention Trial (PPT) is to determine whether a low fat, high fiber, high vegetable and fruit eating plan will decrease the recurrence of adenomatous polyps of the large bowel. Secondary objectives of the PPT include 1) evaluating the effectiveness of the intervention program with respect to participant achievement of dietary goals; 2) examining the relation of dietary change and biochemical markers in blood; and 3) assessing the impact of the intervention on quality of life indicators.

BACKGROUND:

Nearly 60,000 men and women will die from large bowel cancer in the United States this year, making it the second leading cause of death from malignant disease in this country. The evidence that diet plays a key role in large bowel carcinogenesis is strong and growing. The PPT was undertaken because it is unlikely, with respect to diet and large bowel cancer, that any combination of further animal research, clinical investigations employing non-neoplastic endpoints, or observational epidemiologic studies would be sufficiently persuasive to influence public health policy.

A large body of ecologic, analytic epidemiologic, human metabolic, and animal experimental data suggests that three dietary factors increase the risk of large bowel cancer: high dietary fat, low dietary fiber, and low vegetable and fruit intake. Previous dietary intervention studies have generally focused on a single nutrient. The PPT is unique in that three dietary factors are being investigated simultaneously through intervention with a realistic, comprehensive dietary pattern change. NCI investigators adopted this multiple-goal dietary intervention strategy in the PPT for several reasons: people eat foods, not isolated nutrients; there may be unknown protective food constituents not encompassed in a single-nutrient intervention; and there may well be important synergistic effects of various food components best captured in a comprehensive, multifactor dietary pattern. Moreover, by embracing three promising dietary hypotheses simultaneously, the PPT intervention is intended to maximize the possibility of reducing polyp recurrence. The direct demonstration of any effect of diet on the large bowel neoplastic process would be a major advance.

Large bowel adenomas (polyps) present a unique opportunity to conduct an intervention trial because of the high prevalence of these lesions in the general population (over 30% in adults over 50 years of age), the high polyp recurrence rate (at least 10% annually) in those who have undergone adenoma removal, and the strong link between adenomas and cancer (the so-called adenoma-carcinoma sequence). It is generally accepted that large bowel adenomas are an obligate precursor lesion for most large bowel cancers. An intervention reducing the recurrence of large bowel polyps would thus have a strong likelihood of reducing the incidence of large bowel cancer.

DESIGN:

The PPT is a randomized, controlled trial being carried out at eight Clinical Centers in the United States. The Data and Nutrition Coordinating Center (DNCC) is Westat, Inc., Rockville, Maryland. The target sample size of 2000 permits the detection with 90% power of a reduction of 24% in the polyp recurrence rate.

The dietary goals for the intervention arm are 20% of calories from fat, 18g fiber/1000 kcal, and 5-8 servings of fruits and vegetables (the exact number based on caloric intake). The usual (control) diet, based on data from national surveys, is expected to comprise approximately 35% of calories from fat, 10-15 g per day of dietary fiber, and 3.5 servings of vegetables and fruits daily.

The overall strategy for the intervention program is to reduce calories from fat and to replace them with calories from fruits vegetables and grains thus increasing dietary fiber intake. The intervention program, patterned after the approach used in the feasibility phase of the Women's Health Trial, integrates nutrition education and behavior modification techniques. Although initial counseling sessions are carried out one-on-one by the PPT nutritionists, most intervention group members participate in group counseling after the first year.

The control group is not offered a nutrition intervention program since the general strategy adopted for this group will be minimum interference with customary diets while collecting nutritional data considered necessary for appropriate comparison with the nutrition intervention group. Subjects in the control group are expected to maintain their usual diet.

Three different dietary assessment instruments are used in the PPT: a modified Block/NCI Food Frequency Questionnaire (FFQ), Four Day Food Records (4DFR), and 24 Hour Recalls.

Participants undergo colonoscopy again at one (T1) and four (T4) years into the study. Over 280 endoscopists participating in the PPT carry out the T1 and T4 colonoscopies. Although the recurrence of one or more adenomas is the primary endpoint of the study, it will also be possible to relate the dietary intervention to number, size, and histotype of polyps. Because some polyps (10-15%) tend to be missed at baseline, the primary analytic interval (on which sample size calculations were based) is T1 through T4.

The presence of one or more adenomas at the qualifying colonoscopy--a key eligibility factor for PPT--was determined by Clinical Center trial pathologists who had been previously oriented by the central pathologists to PPT pathologic criteria. The number, size, and location of adenomas at baseline was determined by the participating endoscopists. To standardize the histologic diagnoses used in endpoint ascertainment, the PPT requires that histologic type and extent of atypia be determined by the central pathologists for all lesions removed at baseline, T1, and T4.

Blood specimens are collected on all participants annually; these are analyzed on a 20% participant sample (the same individuals for whom the diet records are analyzed) for lipids, carotenoids, and vitamins A and E. Blood specimens are also available for other analyses including hormone and molecular genetic analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women who at the time of randomization are 35 years of age or older and have had removed within 6 months of randomization one or more adenomatous polyps confirmed histologically by the Clinical Center trial pathologist.

EXCLUSION CRITERIA:

Persons with any of the following characteristics are ineligible for the study:

Carcinoma in any polyp removed at baseline endoscopy. High grade dysplasia is not considered carcinoma for purposes of study eligibility.

Failure to examine the cecum during baseline colonoscopy.

Incomplete removal of polyps at baseline colonoscopy.

Surgical removal of polyps.

Familial polyposis or other polyposis syndromes.

Adenomatous polyp discovered before the age of 35.

History of large bowel cancer, including intramucosal carcinoma.

History of histologically or radiographically confirmed inflammatory bowel disease (ulcerative colitis or Crohn's disease).

History of large bowel resection.

Weight move than 150% of desirable weight according to the 1983 Metropolitan Life Insurance Tables.

Use of lipid-lowering drugs in pharmacologic doses in the last month.

Major life-limiting conditions reducing likelihood of completing 4-year follow-up.

Already consuming a dietary pattern similar to the intervention eating plan.

Any dietary practice, behavior, or attitude that would substantially limit adherence to the intervention program.

Participation in other clinical studies that may interfere with participation in the PPT.

Unable or unwilling to sign informed consent form.

Found to be unreliable and uncooperative providers of dietary information during the pre-randomization period.

Able to give reasonable assurance of remaining in the Clinical Center area for duration of the study.

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2079 (Actual)
Dates: Start 1991-06-19 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of polyps in the colon | Yearly for 4 years
  Adenoma recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gwen A Murphy, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hill MJ, Morson BC, Bussey HJ. Aetiology of adenoma--carcinoma sequence in large bowel. Lancet. 1978 Feb 4;1(8058):245-7. doi: 10.1016/s0140-6736(78)90487-7. PMID 74668
- [Background] Zaridze DG. Environmental etiology of large-bowel cancer. J Natl Cancer Inst. 1983 Mar;70(3):389-400. No abstract available. PMID 6300495
- [Background] Drasar BS, Irving D. Environmental factors and cancer of the colon and breast. Br J Cancer. 1973 Feb;27(2):167-72. doi: 10.1038/bjc.1973.20. PMID 4694388
- [Derived] Byrd DA, Vogtmann E, Ortega-Villa AM, Wan Y, Gomez M, Hogue S, Warner A, Zhu B, Dagnall C, Jones K, Hicks B, Albert PS, Murphy G, Sinha R. Prospective and Cross-sectional Associations of the Rectal Tissue Microbiome with Colorectal Adenoma Recurrence. Cancer Epidemiol Biomarkers Prev. 2023 Mar 6;32(3):435-443. doi: 10.1158/1055-9965.EPI-22-0608. PMID 36525653
- [Derived] Perera T, Young MR, Zhang Z, Murphy G, Colburn NH, Lanza E, Hartman TJ, Cross AJ, Bobe G. Identification and monitoring of metabolite markers of dry bean consumption in parallel human and mouse studies. Mol Nutr Food Res. 2015 Apr;59(4):795-806. doi: 10.1002/mnfr.201400847. Epub 2015 Feb 23. PMID 25641932